CLINICAL TRIAL: NCT04454801
Title: Expert Behaviors in Ultrasound Guided Regional Anesthesia A Mixed-Methods Study
Brief Title: Expert Behaviors USGRA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 19-6238
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-06

CONDITIONS: Anesthesia Education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Expert-performance begins by focusing specifically on the end-product of training and experience in the hands of the expert. By defining expert behaviors and techniques, investigators can guide learners and non-expert practitioners by offering them models to emulate. At Toronto Western Hospital (TWH), there are more than ten expert attending regional anesthesiologists who routinely provide clinical patient care in the block room. The primary objective of this study is to qualitatively and quantitatively examine behavior of experts performing ultrasound guided regional anesthesia techniques to identify those which are consistent and unique, and which may underpin expert performance.

ELIGIBILITY:
Inclusion Criteria:

* All elective patients coming to the regional BR at TWH aged 18-80

Exclusion Criteria:

* Any contraindication to USGRA (LA allergy, patient refusal, infection at injection site, etc.)
* Inability to read or speak or comprehend English fluently

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a mixed methods assessment study to be completed at TWH. We will recruit 10 fellowship-trained regional anesthesiology and pain medicine staff anesthesiologists to perform USGRA blocks while being video-recorded. Here, we specifically define expert as a staff anesthesiologist who has completed a fellowship in regional anesthesia and/or chronic pain and has at least 6-years of post-fellowship clinical experience with USGRA.
  Consent will also be sought from 180 patients undergoing USGRA for surgical procedures at TWH to have the block completed by an expert, as previously defined, and to have the procedure recorded.
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2020-08-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Qualitative behaviors of experts performing UGRA techniques during pre-procedural discussion | 1 hour before procedure
  Reviewers will identify behaviors exhibited by the expert operators during pre-procedural discussion
Qualitative behaviors of experts performing UGRA techniques during patient and equipment preparation | 0.5 hour before procedure
  Reviewers will identify behaviors exhibited by the expert operators during patient and equipment preparation
Qualitative behaviours of experts performing UGRA techniques during ultrasound scanning of the target area; | 10 minutes before procedure
  Reviewers will identify behaviors exhibited by the expert operators during ultrasound scanning of the target area;
Qualitative behaviours of experts performing UGRA techniques during needle advancement and local anesthetic deposition around the target nerve(s) | during procedure
  Reviewers will identify behaviors exhibited by the expert operators during needle advancement and local anesthetic deposition around the target nerve(s).
Quantitative data on block effectiveness defined by blocks requiring top-up | 0-1 hour after procedure
  number of top-up will be collected
Quantitative data on block effectiveness defined by blocks requiring conversion to GA | 0-1 hour after procedure
  Incidence will be documented in case conversion to GA is needed
Quantitative data on time to surgical anesthesia | 0-1 hour after procedure
  defined by final needle removal to surgical anesthesia
Quantitative data on time to block completion | 0-1 hour after procedure
  defined by needle insertion to final needle removal

CONTACTS AND LOCATIONS:
Overall Officials: Ki Jinn Chin, MD, Principal Investigator — University Health Network, Toronto